CLINICAL TRIAL: NCT04936165
Title: Circulation and Oxygenation Changes of Deep Tissue Respond on Low Level Light/Laser Therapy (LLLT) in the Healthy Population
Brief Title: Circulation and Oxygenation Changes of Deep Tissue Respond on LLLT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ting Li (Unknown)
Responsible Party: Sponsor-Investigator, Ting Li, Full professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Deep Optical Theranastics
Record Dates: First submitted 2020-11-09; First posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-02

CONDITIONS: Low Level Light/Laser Therapy; Near Infrared Spectroscopy
Keywords: Low level light/laser therapy; Near infrared spectroscopy
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy experimental participants (Experimental): The participants sat in a a quiet and darkened room with the upper arm at heart level and the forearm in an upward angle of 30°, 15-20 min prior to the experiment.
  The experiments consists of 5-min rest, 90s inflated wrist cuff (240 mmHg) with 30s VO(one minute later), 3-min rest, 10-min intervention, the same 4.5-min process of the wrist cuff, VO and rest.
  Device: Optical monitor for hemodynamic parameter. Near infrared spectroscopy probes of tow wavelengths were attached on the participants' forearm and brain to detect the changes of hemodynamic parameters.
  Interventions: Procedure: Low-Level Laser Therapy
- Healthy controlled participants (No Intervention): The participants sat in a a quiet and darkened room with the upper arm at heart level and the forearm in an upward angle of 30°, 15-20 min prior to the experiment.
  The experiments consists of 5-min rest, 90s inflated wrist cuff (240 mmHg) with 30s VO(one minute later), 3-min rest, 10-min rest, the same 4.5-min process of the wrist cuff, VO and rest.
  Device: Optical monitor for hemodynamic parameter. Near infrared spectroscopy probes of tow wavelengths were attached on the participants' forearm and brain to detect the changes of hemodynamic parameters.

INTERVENTIONS:
Procedure: Low-Level Laser Therapy — Use 810-nm-photosource to irradiate the participants' brain and forearm for 10 minutes with a water-cooling radiator to keep it at 25 ± 0.5 ℃.
  Arms: Healthy experimental participants

SUMMARY:
This study aims to investigate the circulation and oxygenation changes of deep tissue respond on low level light/laser therapy (LLLT) in the healthy population. The investigators used a self-made near infrared spectroscopy (NIRS) instrument to noninvasively monitor hemodynamic indicators of brain and forearm muscle groups, including total hemoglobin ([tHb]), and blood flow (BF) and oxygen consumption (VO2).

DETAILED DESCRIPTION:
Low level light/laser therapy (LLLT) employs visible or near-infrared light generated from a laser or light emitting diode (LED) system. It has beneficial effects on a wide range of disease, including improving wound healing, reducing pain, improving memory, treat cancer, and many other human applications. This study aims to investigate the circulation and oxygenation changes of deep tissue respond on low level light/laser therapy (LLLT) in the healthy population. The investigators used a self-made near infrared spectroscopy (NIRS) instrument to noninvasively monitor hemodynamic indicators of brain and forearm muscle groups, including total hemoglobin ([tHb]), and blood flow (BF) and oxygen consumption (VO2). Then the investigators concluded the effect of LLLT, according to compare the difference between the experimental group and control group.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants with no strenuous exercise or alcohol consumption prior to the test

Exclusion Criteria:

* having risk factors associated with cardiovascular disease

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-06-25 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Δ[HbO2] | through study completion, an average of 1 year
  changes of oxyhemoglobin concentration
Δ[Hb] | through study completion, an average of 1 year
  changes of deoxy-hemoglobin concentration
Δ[tHb] | through study completion, an average of 1 year
  changes of total hemoglobin concentration

SECONDARY OUTCOMES:
Subcutaneous fat thickness | through study completion, an average of 1 year
  the subcutaneous fat thickness of the forearm

CONTACTS AND LOCATIONS:
Locations (1):
- NIRS assessment for brain death, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No